CLINICAL TRIAL: NCT04102865
Title: NPWT Pre-registration Study: A Prospective, Multicentre Trial to Assess Performance, Safety and Efficacy of a Single-use NPWT Device
Brief Title: Performance, Safety and Efficacy of NPWT Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CT1705POB
Record Dates: First submitted 2018-04-26; First posted 2019-09-25 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2022-12

CONDITIONS: Wound Healing and Prevention
Keywords: surgical complication; Negative-Pressure Wound Therapy (NPWT); negative pressure; knee arthroplasty; abdominal incision
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominal (Other): Abdominal surgery type with investigational single use NPWT dressing
  Interventions: Device: Negative-Pressure Wound Therapy (NPWT)
- Knee (Other): Knee surgery type with investigational single use NPWT dressing
  Interventions: Device: Negative-Pressure Wound Therapy (NPWT)

INTERVENTIONS:
Device: Negative-Pressure Wound Therapy (NPWT) — Investigational single use disposable negative pressure system. The system is capable of delivering up to 80 mm Hg negative pressure to a wound or surgical incision site and managing low to moderate levels of exudate or fluid generated by the wound or incision. The therapy may be administered for up to 7 days.
  Other Names: NPWT system

SUMMARY:
Smith & Nephew are assessing a new investigational single use NPWT system.

DETAILED DESCRIPTION:
Smith & Nephew are assessing a new investigational single use NPWT system. There is a significant amount of clinical evidence to show that NPWT may reduce oedema, increase healing and reduce chance of infection, through maintenance of pressure therapy, in closed incisions. Subjects with abdominal incisions and knee incisions following knee surgery will be recruited to the study and receive NPWT for 7 days. The performance of the system will be logged by the device and acceptability of the device will be assessed by patient and clinician. Safety will be assessed with a 30 day follow up to assess complications and device related events.

ELIGIBILITY:
Inclusion Criteria:

* The subject must provide written informed consent.
* Subjects eighteen (18) years of age or older.
* Willing and able to make all required study visits.
* Able to follow instructions.
* Subject is suitable to participate in the study in the opinion of the Investigator
* In Orthopaedic surgery: subject is scheduled for an elective primary knee replacement arthroplasty and American Society of Anesthesiologists (ASA) score of 2-3 (Phase 1 only)
* In Abdominal surgery: subject is scheduled for an elective open or laparoscopic gastrointestinal and/or gynaecological surgery with incision ≥5 cm and has an ASA score of 2-3.
* Immediately after the surgery, subject will have one suitable closed abdominal or knee surgery incision (if there is more than one incision, then the clinician should choose the one which, in their opinion, is most suited for Negative Pressure Wound Therapy) that fits under the absorbent dressing area of the appropriate Negative Pressure dressing sizes .

Exclusion Criteria:

* Contraindications (per the Investigator Brochure) or hypersensitivity to the use of the investigational product or their components (e.g. silicone adhesives and polyurethane films [direct contact with incision], acrylic adhesives [direct contact with skin], polyethylene fabrics and super-absorbent powders [polyacrylates]) within the dressing).
* Subjects with extremely fragile skin who require the use of SECURA™ non-sting barrier skin wipes and have hypersensitivity to the ingredients in the wipes
* Participation in the treatment period of another similar clinical trial (wound care related) within thirty (30) days of operative visit or during the study.
* Subjects with skin features (e.g. tattoos, skin colour, pre-existing scarring) which in the opinion of the Investigator, will interfere with the study assessments.
* Subjects attending for an operation at the same surgery site (anatomical location) within the last 3 months
* Subjects undergoing a procedure as part of palliative care (to be confirmed during surgery).
* Subjects where the area of the device would be placed on a load-bearing anatomical location (i.e. areas vulnerable to pressure damage).
* Subjects with incisions that are actively bleeding unless haemostasis has been achieved (to be confirmed during surgery).
* Subjects with infected skin lesions or incisions at the time of surgery (any area of the body).
* Subjects who have participated previously in this clinical trial
* Subjects with a history of poor compliance with medical treatment.
* Subjects with a BMI ≥ 40.
* Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jeffery, Principal Investigator — Queen Elizabeth Hospital, Birmingham, UK
Locations (8):
- United Kingdom (8):
  - Worthing Hospital, Worthing, West Sussex
  - Queen Elizabeth Hospital, Birmingham
  - Western General Hospital, Edinburgh
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - North Tyneside General Hospital, North Shields
  - RJAH Orthopaedic Hospital, Oswestry
  - Peterborough City Hospital, Peterborough
  - Torbay Hospital, Torquay

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began 12 July 2019 to 01 February 2022 across 8 investigative sites.
Period: Overall Study
Arm/Group | Abdominal | Knee
Started | 68 | 22
Completed | 61 | 22
Not Completed | 7 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population utilized. Participants with Intent-to-Treat (ITT) that included all enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdominal | Knee | Total
Number analyzed (Participants) | 68 | 22 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (11.9) | 70.4 (7.6) | 67.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 40
  Male | 42 | 8 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 67 | 22 | 89
  Race: Asian | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White British | 63 | 22 | 85
  Ethnicity: White Irish | 1 | 0 | 1
  Ethnicity: Any Other White Background | 2 | 0 | 2
  Ethnicity: White and Asian Mixed | 1 | 0 | 1
  Ethnicity: Not Stated | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 68 | 22 | 90
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (5.2) | 31.5 (3.4) | 28.9 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Negative Pressure Maintenance at Nominal 80 mmHg
Description: Negative pressure maintenance at nominal 80 mmHg assessed as the average of the negative pressure values recorded by the device for Abdominal and Knee surgery types. This data was summarized to show an average negative pressure provided over the treatment duration.
Time Frame: 30 days post-op
Population: Full Analysis Set (FAS) population included enrolled participants with available data for the surgery type specified.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 58 | 18
millimeters of mercury (mmHg) | -71.5 (25.1) | -56.0 (28.2)

2. Primary Outcome: Dressing Wear Time
Description: Dressing wear time in days as assessed of any unplanned dressing change by Abdominal and Knee surgery type.
Time Frame: 7 days
Population: Full Analysis Set (FAS) population included enrolled participants with available data for the surgery type specified.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 68 | 22
days | 5.7 (2.4) | 5.3 (2.1)

3. Primary Outcome: Exudate Management (Occurrence of Exudate Leaks)
Description: Number of participants with occurrence of exudate leaks. Leakage classified as 'Any Leak' (Yes/No) by Abdominal and Knee surgery type.
Time Frame: 7 days
Population: Full Analysis Set (FAS) population included enrolled participants with available data for the surgery type specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 68 | 22
Participants
  Any Leak: Yes | 5 | 12
  Any Leak: No | 63 | 10

4. Secondary Outcome: Incidence of Surgical Site Infection (SSI)
Description: Number of participants with incidence of Surgical Site Infection (SSI) within 30 days of surgery classified using Centers for Decease Control (CDC) criteria of:
  * Superficial Infection
  * Deep Infection
  * Organ Space Infection
  * Other
Time Frame: 30 days
Population: Full Analysis Set (FAS) population included all enrolled participants with available data for the specified assessment. Out of 90 (68 Abdominal, 22 Knee) participants overall, 5 (5 Abdominal, 0 Knee) participants experienced at least one Surgical Site Infection (SSI) indicated by the given criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 68 | 22
Participants
  Superficial Infection | 3 | 0
  Deep Infection | 2 | 0
  Organ Space Infection | 1 | 0
  Other | 1 | 0

5. Secondary Outcome: Incidence of Surgical Site Complications (SSC)
Description: Number of participants with incidence of Surgical Site Complications (SSC) within 30 days of surgery categorized as:
  * Deep Dehiscence
  * Superficial Dehiscence
  * Partial Dehiscence
  * Total Dehiscence
  * Seroma
  * Necrosis
  * Hematoma
  * Suture Abscess
  * Other
Time Frame: 30 days
Population: Full Analysis Set (FAS) population included all enrolled participants with available data for the specified assessment. Out of 90 (68 Abdominal, 22 Knee) participants overall, 10 (9 Abdominal, 1 Knee) participants experienced at least one Surgical Site Complication (SSC) indicated by the given criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 68 | 22
Participants
  Deep Dehiscence | 2 | 0
  Superficial Dehiscence | 6 | 0
  Partial Dehiscence | 5 | 0
  Total Dehiscence | 1 | 0
  Seroma | 0 | 0
  Necrosis | 0 | 0
  Haematoma | 2 | 0
  Suture Abscess | 0 | 0
  Other | 2 | 1

6. Secondary Outcome: Condition of Peri-Wound Skin Assessed Through Visual Inspection
Description: Condition of peri-wound skin assessed through visual inspection by the investigator at baseline, 7, 14, and 30 days. Number of participants by Abdominal and Knee surgery type where skin was categorized with any condition that applied (i.e., multiple selections possible) from the following criteria:
  * Healthy
  * Fragile
  * Inflamed
  * Erythema
  * Bruising
  * Eczematous
  * Dry and Flaky
  * Macerated
  * Other
Time Frame: Baseline, 7 days, 14 days, and 30 days
Population: Full Analysis Set (FAS) population included enrolled participants with available data for the specified assessment at the time point indicated. Because multiple responses were possible, "Healthy" skin could be recorded along with any other conditions. Where this occurred, the investigator believed the other condition(s) selected did not affect the healthiness of the skin.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 68 | 22
Participants
  Baseline: Healthy | 68 | 22
  Baseline: Fragile | 4 | 0
  Baseline: Inflamed | 2 | 0
  Baseline: Erythema | 2 | 0
  Baseline: Bruising | 0 | 1
  Baseline: Eczematous | 0 | 0
  Baseline: Dry and Flaky | 0 | 0
  Baseline: Macerated | 0 | 0
  Baseline: Other | 1 | 0
  7 Days: Healthy: number analyzed (Participants) | 64 | 19
  7 Days: Healthy | 59 | 19
  7 Days: Fragile: number analyzed (Participants) | 64 | 19
  7 Days: Fragile | 1 | 0
  7 Days: Inflamed: number analyzed (Participants) | 64 | 19
  7 Days: Inflamed | 4 | 2
  7 Days: Erythema: number analyzed (Participants) | 64 | 19
  7 Days: Erythema | 2 | 1
  7 Days: Bruising: number analyzed (Participants) | 64 | 19
  7 Days: Bruising | 35 | 12
  7 Days: Eczematous: number analyzed (Participants) | 64 | 19
  7 Days: Eczematous | 1 | 0
  7 Days: Dry and Flaky: number analyzed (Participants) | 64 | 19
  7 Days: Dry and Flaky | 3 | 1
  7 Days: Macerated: number analyzed (Participants) | 64 | 19
  7 Days: Macerated | 1 | 0
  7 Days: Other: number analyzed (Participants) | 64 | 19
  7 Days: Other | 4 | 3
  14 Days: Healthy: number analyzed (Participants) | 64 | 21
  14 Days: Healthy | 59 | 21
  14 Days: Fragile: number analyzed (Participants) | 64 | 21
  14 Days: Fragile | 2 | 0
  14 Days: Inflamed: number analyzed (Participants) | 64 | 21
  14 Days: Inflamed | 7 | 3
  14 Days: Erythema: number analyzed (Participants) | 64 | 21
  14 Days: Erythema | 9 | 2
  14 Days: Bruising: number analyzed (Participants) | 64 | 21
  14 Days: Bruising | 17 | 5
  14 Days: Eczematous: number analyzed (Participants) | 64 | 21
  14 Days: Eczematous | 2 | 0
  14 Days: Dry and Flaky: number analyzed (Participants) | 64 | 21
  14 Days: Dry and Flaky | 5 | 0
  14 Days: Macerated: number analyzed (Participants) | 64 | 21
  14 Days: Macerated | 1 | 0
  14 Days: Other: number analyzed (Participants) | 64 | 21
  14 Days: Other | 6 | 3
  30 Days: Healthy: number analyzed (Participants) | 61 | 22
  30 Days: Healthy | 59 | 22
  30 Days: Fragile: number analyzed (Participants) | 61 | 22
  30 Days: Fragile | 4 | 0
  30 Days: Inflamed: number analyzed (Participants) | 61 | 22
  30 Days: Inflamed | 3 | 1
  30 Days: Erythema: number analyzed (Participants) | 61 | 22
  30 Days: Erythema | 3 | 0
  30 Days: Bruising: number analyzed (Participants) | 61 | 22
  30 Days: Bruising | 0 | 2
  30 Days: Eczematous: number analyzed (Participants) | 61 | 22
  30 Days: Eczematous | 1 | 0
  30 Days: Dry and Flaky: number analyzed (Participants) | 61 | 22
  30 Days: Dry and Flaky | 9 | 4
  30 Days: Macerated: number analyzed (Participants) | 61 | 22
  30 Days: Macerated | 0 | 0
  30 Days: Other: number analyzed (Participants) | 61 | 22
  30 Days: Other | 4 | 2

7. Secondary Outcome: Condition of Skin Under the Investigative Single Use Negative-Pressure Wound Therapy (NPWT) Dressing Assessed Through Visual Inspection
Description: Condition of skin under investigative single use Negative-Pressure Wound Therapy (NPWT) dressing assessed through visual inspection by the investigator at baseline, 7, 14, and 30 days. Number of participants by Abdominal and Knee surgery type where skin was categorized with any condition that applied (i.e., multiple selections possible) from the following criteria:
  * Healthy
  * Fragile
  * Inflamed
  * Erythema
  * Bruising
  * Eczematous
  * Dry and Flaky
  * Macerated
  * Other
Time Frame: Baseline, 7 days, 14 days, and 30 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 68 | 22
Participants
  Baseline: Healthy | 68 | 22
  Baseline: Fragile | 1 | 0
  Baseline: Inflamed | 0 | 0
  Baseline: Erythema | 0 | 0
  Baseline: Bruising | 13 | 0
  Baseline: Eczematous | 0 | 0
  Baseline: Dry and Flaky | 0 | 0
  Baseline: Macerated | 0 | 0
  Baseline: Other | 0 | 0
  7 Days: Healthy: number analyzed (Participants) | 64 | 19
  7 Days: Healthy | 62 | 19
  7 Days: Fragile: number analyzed (Participants) | 64 | 19
  7 Days: Fragile | 0 | 0
  7 Days: Inflamed: number analyzed (Participants) | 64 | 19
  7 Days: Inflamed | 1 | 0
  7 Days: Erythema: number analyzed (Participants) | 64 | 19
  7 Days: Erythema | 1 | 0
  7 Days: Bruising: number analyzed (Participants) | 64 | 19
  7 Days: Bruising | 10 | 3
  7 Days: Eczematous: number analyzed (Participants) | 64 | 19
  7 Days: Eczematous | 0 | 0
  7 Days: Dry and Flaky: number analyzed (Participants) | 64 | 19
  7 Days: Dry and Flaky | 1 | 0
  7 Days: Macerated: number analyzed (Participants) | 64 | 19
  7 Days: Macerated | 0 | 0
  7 Days: Other: number analyzed (Participants) | 64 | 19
  7 Days: Other | 3 | 3
  14 Days: Healthy: number analyzed (Participants) | 64 | 21
  14 Days: Healthy | 64 | 21
  14 Days: Fragile: number analyzed (Participants) | 64 | 21
  14 Days: Fragile | 2 | 0
  14 Days: Inflamed: number analyzed (Participants) | 64 | 21
  14 Days: Inflamed | 1 | 1
  14 Days: Erythema: number analyzed (Participants) | 64 | 21
  14 Days: Erythema | 1 | 0
  14 Days: Bruising: number analyzed (Participants) | 64 | 21
  14 Days: Bruising | 6 | 0
  14 Days: Eczematous: number analyzed (Participants) | 64 | 21
  14 Days: Eczematous | 1 | 0
  14 Days: Dry and Flaky: number analyzed (Participants) | 64 | 21
  14 Days: Dry and Flaky | 1 | 1
  14 Days: Macerated: number analyzed (Participants) | 64 | 21
  14 Days: Macerated | 0 | 0
  14 Days: Other: number analyzed (Participants) | 64 | 21
  14 Days: Other | 2 | 0
  30 Days: Healthy: number analyzed (Participants) | 61 | 21
  30 Days: Healthy | 60 | 21
  30 Days: Fragile: number analyzed (Participants) | 61 | 21
  30 Days: Fragile | 1 | 0
  30 Days: Inflamed: number analyzed (Participants) | 61 | 21
  30 Days: Inflamed | 1 | 0
  30 Days: Erythema: number analyzed (Participants) | 61 | 21
  30 Days: Erythema | 3 | 0
  30 Days: Bruising: number analyzed (Participants) | 61 | 21
  30 Days: Bruising | 0 | 0
  30 Days: Eczematous: number analyzed (Participants) | 61 | 21
  30 Days: Eczematous | 1 | 0
  30 Days: Dry and Flaky: number analyzed (Participants) | 61 | 21
  30 Days: Dry and Flaky | 3 | 0
  30 Days: Macerated: number analyzed (Participants) | 61 | 21
  30 Days: Macerated | 0 | 0
  30 Days: Other: number analyzed (Participants) | 61 | 21
  30 Days: Other | 1 | 0

8. Secondary Outcome: Wound and Skin Visual Analog Scale (VAS) Score Assessment
Description: Wound and Skin VAS score assessment at 7, 14 and 30 days. Scores range from 0 to 100 with a low score associated to a wound with a major gapping, dehiscence, severe inflammation and/or infection (i.e., poor outcome); and a high correspond to a completely healed wound with no evidence for inflammation (i.e., excellent outcome).
Time Frame: 7 days, 14 days, and 30 days
Population: Full Analysis Set (FAS) population included enrolled participants with available data for the specified assessment at the time point indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 66 | 22
score on a scale
  7 Days: number analyzed (Participants) | 63 | 19
  7 Days | 79.0 (26.7) | 89.9 (7.4)
  14 Days: number analyzed (Participants) | 65 | 21
  14 Days | 81.4 (26.1) | 89.4 (10.4)
  30 Days | 85.0 (27.6) | 95.0 (5.6)

9. Secondary Outcome: Range of Motion Assessment (ROM) for the Knee
Description: Range of Motion (ROM) assessment for the knee at pre-operative visit, post-operative visit, 7, 14 and 30 days.
Time Frame: 30 days
Population: Data reported for knee extension in Knee Group interpreted as negative (extension deficit) or positive (actual extension). Therefore, ROM can be the sum or difference of reported knee flexion & extension. Because different Investigators applied different interpretations, there is low confidence in reliability of ROM data. Further investigation is required with additional clinical evaluations before the investigational NPWT device can be considered suitable for consideration in TKA subjects.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Knee
Number analyzed (Participants) | 22
degrees
  Pre-Operative - Flexion | 102.5 (17.2)
  Pre-Operative - Extension Angle | 9.4 (7.7)
  Pre-Operative - ROM | 93.1 (20.7)
  Post-Operative - Flexion: number analyzed (Participants) | 20
  Post-Operative - Flexion | 61.6 (20.3)
  Post-Operative - Extension Angle: number analyzed (Participants) | 21
  Post-Operative - Extension Angle | 6.6 (5.9)
  Post-Operative - ROM: number analyzed (Participants) | 20
  Post-Operative - ROM | 54.9 (21.6)
  Day 7 (Pre-Dressing Removal) - Flexion: number analyzed (Participants) | 15
  Day 7 (Pre-Dressing Removal) - Flexion | 75.5 (16.1)
  Day 7 (Pre-Dressing Removal) - Extension Angle: number analyzed (Participants) | 14
  Day 7 (Pre-Dressing Removal) - Extension Angle | 14.2 (9.5)
  Day 7 (Pre-Dressing Removal) - ROM: number analyzed (Participants) | 14
  Day 7 (Pre-Dressing Removal) - ROM | 61.6 (16.6)
  Day 7 (Post-Dressing Removal) - Flexion: number analyzed (Participants) | 19
  Day 7 (Post-Dressing Removal) - Flexion | 75.6 (19.7)
  Day 7 (Post-Dressing Removal) - Extension Angle: number analyzed (Participants) | 19
  Day 7 (Post-Dressing Removal) - Extension Angle | 11.2 (6.9)
  Day 7 (Post-Dressing Removal) - ROM: number analyzed (Participants) | 19
  Day 7 (Post-Dressing Removal) - ROM | 64.4 (18.2)
  Day 14 - Flexion: number analyzed (Participants) | 21
  Day 14 - Flexion | 86.3 (17.2)
  Day 14 - Extension Angle: number analyzed (Participants) | 21
  Day 14 - Extension Angle | 10.2 (6.3)
  Day 14 - ROM: number analyzed (Participants) | 21
  Day 14 - ROM | 76.0 (18.1)
  Day 30 - Flexion | 100.4 (15.8)
  Day 30 - Extension Angle | 8.7 (5.6)
  Day 30 - ROM | 91.6 (15.9)

10. Secondary Outcome: Level of Pain During Wear of the Investigational Single Use Negative-Pressure Wound Therapy (NPWT) Dressing Assessed by VAS Score
Description: Level of pain during wear by investigational single use Negative-Pressure Wound Therapy (NPWT) Dressing at day 4 and day 7 assessed using a Visual Analog Scale (VAS) from 0 to 100 where a score of 0 indicated no pain and 100 indicated maximum pain.
Time Frame: 4 days and 7 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 60 | 17
score on a scale
  4 Days: number analyzed (Participants) | 59 | 17
  4 Days | 20.2 (24.7) | 41.8 (28.8)
  7 Days | 14.2 (20.5) | 35.4 (26.0)

11. Secondary Outcome: Level of Pain at Dressing Removal of the Investigative Single Use Negative-Pressure Wound Therapy (NPWT) Dressing Assessed by VAS Score
Description: Level of pain during dressing removal by Abdominal and Knee surgery type at treatment discontinuation (up to day 7) assessed using a Visual Analog Scale (VAS) from 0 to 100 where a score of 0 indicated no pain and 100 indicated maximum pain.
Time Frame: 7 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abdominal | Knee
Number analyzed (Participants) | 67 | 22
score on a scale | 12.6 (18.3) | 31.6 (30.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected upon investigational single use NPWT dressing application to 30 days post-surgery.
Arm/Group | Abdominal | Knee
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/22
Serious Adverse Events (participants affected / at risk) | 19/68 | 1/22
Other Adverse Events (participants affected / at risk) | 45/68 | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal (N=68) | Knee (N=22)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Wound haemmorhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pumonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anastomic leak (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) — 2 abdominal subjects discontinued from study due to Serious Adverse Event (SAE)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Application site vesicles (General disorders) | 0 (0) | 1 (1) — Possibly related to study device and study procedure
Dysponea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0) — Subject discontinued from study due to SAE
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal (N=68) | Knee (N=22)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 19 (23) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1)
Application site vesicles (General disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Blood glucose decreased (Investigations) | 1 (2) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 2 (2) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Bloody discharge (Vascular disorders) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Drain site complication (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (4) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Instillation site rash (General disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 7 (8) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lethargic (Nervous system disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Malaise (General disorders) | 3 (6) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasogastric output abnormal (Investigations) | 1 (1) | 0 (0)
Nasogastric output high (Investigations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (24) | 5 (6)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 4 (6) | 0 (0)
Pain (General disorders) | 10 (19) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (2) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postoperative hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 7 (8) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 5 (6) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (14) | 2 (2)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The investigational single use NPWT dressing under investigation within this clinical study has not been submitted for approval and clearance as a medical device within any country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon completion of the Clinical Investigation the PI may prepare the data derived from the Clinical Investigation for publication. Such data will be submitted to the Sponsor for review and comment prior to publication. In order to ensure that Sponsor will be able to make comment and suggestions where pertinent, the material for public dissemination will be submitted for review at least 60 days prior to submission for publication, public dissemination or review by a publication committee.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT04102865/Prot_SAP_000.pdf